CLINICAL TRIAL: NCT03871946
Title: Fibromyalgia in Patient With Impaired Fasting Glucose
Status: Completed | Type: Observational
Sponsor: Hitit University (Other)
Collaborators: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ayla Cagliyan Turk, Principal Investigator, Hitit University
Other Study IDs: Hitit University
Record Dates: First submitted 2019-03-01; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Experimental group subjects with impaired fasting glucose (IFG) (Group 1) underwent an oral glucose tolerance test (OGTT), and patients with levels > 140 mg/dL at the 2nd hour were excluded because they were diagnosed with "impaired glucose tolerance"
  Interventions: Diagnostic Test: oral glucose tolerance test (OGTT)
- control group: The control group (Group 2) comprised 73 patients whose fasting blood glucose level was <100 mg/dL and who agreed to participate in the study.
  Interventions: Diagnostic Test: oral glucose tolerance test (OGTT)

INTERVENTIONS:
Diagnostic Test: oral glucose tolerance test (OGTT) — Implementation of OGTT: The patient was seated in a quiet room after 10-12 h of overnight fasting, and blood samples were drawn. Thereafter, 75 g glucose solution dissolved in 300 mL of water was administeredwithin 5 min. Two hours after this,another blood sample was drawn. During the test, the patient wasn't allowed to rest and eat, but not smoke.

SUMMARY:
To assess the frequency of fibromyalgia among women with impaired fasting glucose.

DETAILED DESCRIPTION:
Objective: To assess the frequency of fibromyalgia among women with impaired fasting glucose.

Materials and Methods: The sample was selected from the patients who applied to the Internal Medicine clinic and whose fasting blood glucose level were ≥100 and <126 mg/dL in their routine examination [Group1 ] and patients whose fasting blood glucose were less than 100 constituted the control group [Group2 ]. Oral glucose tolerance test [OGTT ] has been applied to patients with impaired fasting glucose and whose 2nd hour OGTT levels were under 140 has been included. Patients were evaluated in terms of fibromyalgia according to modified 2010 ACR Fibromiyalgia Criteria. Functional status was assessed by using the Fibromyalgia Impact Questionnaire [FIQ ].

ELIGIBILITY:
Inclusion Criteria:

* the study group subjects: fasting blood glucose level was between 100 and 126 mg/dL;
* the control group subjects: fasting blood glucose level was < 100 mg/dL.

Exclusion Criteria:

* Patients with a severe systemic disease (chronic kidney disease, liver disease etc. ),
* psychiatric disease,
* hypothyroidism or hyperthyroidism,
* any connective tissue disease
* patients who used medications that influenced the fibromyalgia symptoms, such as analgesics, antidepressants, and anticonvulsive medications

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18-65 years female patients
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
the frequency of fibromyalgia among women with impaired fasting glucose. | 16 month
  Moreover, a significantly higher proportion of Group 1 patients (26%, n = 19) than Group 2 patients (11%, n = 8) were diagnosed with FM

IPD SHARING:
Plan to Share IPD: No